CLINICAL TRIAL: NCT05477394
Title: Metabolic Syndrome as a Prognostic Factor for Outcome of Sever SARS-COV-2 Cases.
Brief Title: Metabolic Syndrome as Prognostic Factor for Outcome of Sever SARS-COV-2 Cases.
Acronym: COVID19
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: obsevational
Record Dates: First submitted 2022-03-15; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
SARS-COV-2 crisis is a severe public health concern in the world. It is now well recognized that older age, diabetes mellitus, obesity (BMI > 30 kg/m2), and hypertension increase the risk of complications and death in SARS-COV-2 patients.

This study will describe the spectrum of clinical features, the likely pathophysiologic mechanisms, and potential implications for the management of metabolic syndrome in SARS-COV-2 patients.

DETAILED DESCRIPTION:
SARS-COV-2 (Coronavirus Disease-2019), a disease caused by the coronavirus. SARS-CoV-2 (Sever Acute Respiratory Syndrome-Coronavirus-2) has emerged as a rapidly spreading communicable disease affecting more than 100 countries across the globe at present.

The disease is primarily spread through large respiratory droplets, though the possibility of other routes of transmission cannot be ruled out, as the virus has been found in stool and urine of affected individuals.

The disease severity has varied from mild self-limiting flu-like illness to fulminant pneumonia, respiratory failure and death. Several risk groups have been identified as being at higher risk of developing a more severe form of the disease and, subsequently, have higher mortality. In particular, cardiovascular diseases, hypertension, chronic respiratory diseases, metabolic syndrome (MS), and diabetes mellitus (DM) appear to play an important role in developing a more severe form of the disease with several complications.

Metabolic syndrome is a constellation of cardiovascular risk factors that include abdominal obesity, elevated blood pressure, dysglycemia, atherogenic dyslipidemia, pro-thrombotic state, and pro-inflammatory state).

Clinically, metabolic syndrome is defined as the presence of 3 or more of the following factors: increased waist circumference (population and country-specific cutoff), hypertriglyceridemia (>150 mg/dL or on treatment for hypertriglyceridemia), elevated blood pressure (systolic . 130 and/or diastolic . 85 mm Hg or with a history of hypertension on treatment), reduced high-density lipoprotein cholesterol (<40 mg/dL in males; <50 mg/dL in females), and dysglycemia (.100 mg/dL or on treatment for hyperglycemia)

. Components of metabolic syndrome such as hypertension, type 2 diabetes mellitus (T2DM), and obesity are highly prevalent and significantly increase the risk of hospitalization and mortality in SARS-COV-2 patients.

The pathophysiologic mechanisms for these observations have not been fully explained. A critical interaction between SARS-CoV-2 and the angiotensin-converting enzyme 2 (ACE2) facilitates viral entry into the host cell. ACE2 is expressed in pancreatic islets, vascular endothelium, and adipose tissue, and the SARS-CoV-2 -ACE2 interaction in these tissues, along with other factors governs the spectrum and the severity of clinical manifestations among SARS-COV-2 patients with metabolic syndrome.

Moreover, the pro-inflammatory milieu observed in patients with metabolic syndrome may contribute toward SARS-COV-2-mediated host immune dysregulation, including suboptimal immune responses, hyper inflammation, micro-vascular dysfunction, and thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to for Sever Pneumonic COVID-19 infection with a confirmed positive RT-PCR for COVID-19 and chest computed tomography that is divided into two groups.
* Group one is critical COVID patients with metabolic syndrome .
* Group two is critical COVID without metabolic syndrome .

  1. Age 21-50 years old.
  2. Sex both sexes.
  3. Patients having metabolic syndrome defined before who have:
* Diabetes mellitus.
* Hypertension.
* Obesity( BMI < 30 kg/m2)

Exclusion Criteria:

* 1. Patients below 21 years old. 2. Psychiatric disorders. 3. Lack of consent.

Age Groups: Child, Adult, Older Adult
Study Population: • critical SARS-COV-2 patients.
  * patients admitted to for Sever Pneumonic COVID-19 infection with a confirmed positive RT-PCR for COVID-19 and chest computed tomography that is divided into two groups.
  * Group one is critical COVID patients with metabolic syndrome .
  * Group two is critical COVID witout metabolic syndrome .
  Sample Size: 45 patients for each group
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
The period of time that Covid patients spent in intensive care and its outcome. | 6 months
  We note whether metabolic syndrome in cases of Covid is related to the length of stay in the hospital or not.

SECONDARY OUTCOMES:
number of Covid patients who needed mechanical ventilation. | 6 months
  We note whether metabolic syndrome in cases of Covid is related to the need of mechanical ventilation or not.

CONTACTS AND LOCATIONS:
Overall Officials: amr mo hilal, Study Director — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
we will share data which prove that covid patient with metabolic syndrome has a bad prognosis during his treatment
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 6 months
Access Criteria: send to DR.heba992@gmail.com
URL: http://dr.heba992@gmail.com